CLINICAL TRIAL: NCT01969227
Title: The Effects of Subanesthetic Ketamine on Respiratory Stimulation and Transpulmonary Pressures in Mechanically Ventilated Critically Ill Patients
Brief Title: The Effects of Ketamine on Respiratory Stimulation and Transpulmonary Pressures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Medical Director, Respiratory Care, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001690
Record Dates: First submitted 2013-10-08; First posted 2013-10-25 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation; Airway Patency; Respiratory Depression
Keywords: Subanesthetic ketamine; Mechanical ventilation; Transpulmonary pressure; Spontaneous breathing trial; Extubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental): Adult mechanically ventilated patients who are deemed eligible for a spontaneous breathing trial and are candidates to receive subanesthetic ketamine by the primary critical care team.
  Interventions: Drug: Subanesthetic ketamine

INTERVENTIONS:
Drug: Subanesthetic ketamine — Ketamine drip at a subanesthetic infusion rate (low dose ketamine 5 - 10 mcg/kg/min)

SUMMARY:
Impairment of airway patency is a common cause of extubation failure and opioids and hypnotics can adversely affect airway patency. Ketamine, a noncompetitive antagonist of N-methyl-D-aspartate (NMDA), unlike other anesthetics activates respiratory effort and promotes bronchodilation. At subanesthetic plasma concentration, ketamine reduces both opioid and propofol requirements.

The purpose of this pharmaco-physiological interaction trial is to evaluate the effects of ketamine on breathing and electroencephalography in mechanically ventilated patients.

DETAILED DESCRIPTION:
Maintaining the patency of the upper airway in sedated and anesthetized patients is challenging especially when patients are ready to be weaned from mechanical ventilation. Spontaneous breathing trial (SBT) is used to expedite the weaning process, which oftentimes requires the reduction and/or discontinuation of sedatives and analgesics. In some surgical patients, reducing these medications can lead to pain associated agitation and inability to conduct SBTs, which may prolong the need for mechanical ventilation. Using medications with narcotic sparing effects and that do not cause respiratory depression may allow for the reduction or discontinuation of agents that depress respiratory drive and subsequently facilitate extubation.

Ketamine has been used for many years in critically ill patients for sedation and analgesia. This noncompetitive antagonist of N-methyl-D-aspartate (NMDA) is used as an anesthetic and analgesic and has been shown to reduce opioid consumption and to prevent the development of opioid tolerance. Unlike other anesthetics, ketamine activates respiratory effort and promotes bronchodilation. At subanesthetic plasma concentration, ketamine reduces both opioid and propofol requirements.

The goal of this pharmaco-physiological interaction trial is to evaluate the effects of ketamine at a subanesthetic dose on breathing and electroencephalography. The investigators hypothesize that ketamine drip at a subanesthetic infusion rate (low dose ketamine 5 - 10 mcg/kg/min) is associated with respiratory stimulating effects and does not markedly increase transpulmonary pressure in mechanically ventilated patients.

The primary outcome is respiratory function, assessed through peak inspiratory flow, tidal volume,respiratory rate, duty cycle, and minute ventilation measured 15 minutes prior to initiation of ketamine infusion (to serve as baseline), at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, at which point the infusion is stopped for 3 hours for a final set of measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years admitted to ICU requiring mechanical ventilation
* Suitable for spontaneous breathing trial
* Candidate to received low dose ketamine by the primary critical care team

Exclusion Criteria:

* Esophageal injury
* Allergic to ketamine
* Known neurodegenerative disorders
* Major neurologic disorders (elevated ICP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in peak inspiratory flow | Measured 15 minutes prior to initiation of ketamine infusion, at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, and at 2 hours after stopping the infusion
  Measured using a pneumotach (Hans Rudolph Inc., Shawnee, KS) connected to the ventilation tubing of the patient during the spontaneous breathing trials.
Change in tidal volume | Measured 15 minutes prior to initiation of ketamine infusion, at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, and at 2 hours after stopping the infusion
  Measured using a pneumotach (Hans Rudolph Inc., Shawnee, KS) connected to the ventilation tubing of the patient during the spontaneous breathing trials.
Change in duty cycle | Measured 15 minutes prior to initiation of ketamine infusion, at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, and at 2 hours after stopping the infusion
  Measured using a pneumotach (Hans Rudolph Inc., Shawnee, KS) connected to the ventilation tubing of the patient during the spontaneous breathing trials.
Change in respiratory rate | Measured 15 minutes prior to initiation of ketamine infusion, at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, and at 2 hours after stopping the infusion
  Measured using a pneumotach (Hans Rudolph Inc., Shawnee, KS) connected to the ventilation tubing of the patient during the spontaneous breathing trials.
Change in minute ventilation | Measured 15 minutes prior to initiation of ketamine infusion, at 60 minutes of ketamine infusion at 5mcg/kg/min, at another 60 minutes of infusion at 10mcg/kg/min, and at 2 hours after stopping the infusion
  Measured using a pneumotach (Hans Rudolph Inc., Shawnee, KS) connected to the ventilation tubing of the patient during the spontaneous breathing trials.

SECONDARY OUTCOMES:
Transpulmonary pressure | Continuously throughout the study until stopping the ketamine infusion.
  Standard nutritional nasogastric tube with an integrated esophageal balloon will be inserted if not already in place by a trained physician or respiratory therapist prior to initiation of ketamine drip and will be used for measurement of transpulmonary pressure. for the study period (approximately 5 hours)
Changes in power spectrum densities | Continuously throughout the ketamine infusion until 3 hours after stopping the ketamine infusion.
  Electroencephalography (EEG)-based power spectrum densities will be measured using the Sedline brain function monitor (Masimo Corporation, Irvine, CA)
Oxygen blood saturation | Continuously throughout the ketamine infusion until 3 hours after stopping the ketamine infusion.
  Pulse oxymetry
Changes in volumetric capnography | Periods of at least five minutes during steady state breathing before and after administration of ketamine.
  Measures through volumetric capnography: NICO© device from Respironics (Hartford, CT).
Total narcotic consumption | 3 hours after stopping the ketamine infusion
  Obtained from the medical record and flow sheets.
Number of days mechanically ventilated | 3 hours after stopping the ketamine infusion
  Difference in days between intubation and extubation. Obtained from the medical record and flow sheets.
Richmond Agitation Sedation Scale (RASS) | 3 hours after stopping the ketamine infusion
  Obtained from the medical record and flow sheets.
Critical care pain observation tool (CPOT) | 3 hours after stopping the ketamine infusion
  Obtained from the medical record and flow sheets.
Confusion Assessment Measurement for the ICU (CAM-ICU) | 3 hours after stopping the ketamine infusion
  Obtained from the medical record and flow sheets.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital; Matthias Eikermann, MD, PhD, Study Director — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Eikermann M, Grosse-Sundrup M, Zaremba S, Henry ME, Bittner EA, Hoffmann U, Chamberlin NL. Ketamine activates breathing and abolishes the coupling between loss of consciousness and upper airway dilator muscle dysfunction. Anesthesiology. 2012 Jan;116(1):35-46. doi: 10.1097/ALN.0b013e31823d010a. PMID 22108392
- [Background] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Background] Menigaux C, Fletcher D, Dupont X, Guignard B, Guirimand F, Chauvin M. The benefits of intraoperative small-dose ketamine on postoperative pain after anterior cruciate ligament repair. Anesth Analg. 2000 Jan;90(1):129-35. doi: 10.1097/00000539-200001000-00029. PMID 10624993
- [Background] Hirota K, Hashimoto Y, Sakai T, Sato T, Ishihara H, Matsuki A. In vivo spasmolytic effect of ketamine and adrenaline on histamine-induced airway constriction. Direct visualization method with a superfine fibreoptic bronchoscope. Acta Anaesthesiol Scand. 1998 Feb;42(2):184-8. doi: 10.1111/j.1399-6576.1998.tb05106.x. PMID 9509200
- [Background] Morel DR, Forster A, Gemperle M. Noninvasive evaluation of breathing pattern and thoraco-abdominal motion following the infusion of ketamine or droperidol in humans. Anesthesiology. 1986 Oct;65(4):392-8. doi: 10.1097/00000542-198610000-00008. PMID 3767037
- [Background] Kissin I, Bright CA, Bradley EL Jr. The effect of ketamine on opioid-induced acute tolerance: can it explain reduction of opioid consumption with ketamine-opioid analgesic combinations? Anesth Analg. 2000 Dec;91(6):1483-8. doi: 10.1097/00000539-200012000-00035. PMID 11094005